CLINICAL TRIAL: NCT00484939
Title: A Randomised, Open-label Phase III Study to Assess Efficacy and Safety of Bevacizumab in Combination With Capecitabine as First-line Treatment for Elderly Patients With Metastatic Colorectal Cancer
Brief Title: A Study of Bevacizumab (Avastin) in Combination With Capecitabine (Xeloda) in Elderly Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO19286
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Results first posted 2014-06-10 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Capecitabine

ARMS (2):
- Bevacizumab + capecitabine (Experimental): Participants received bevacizumab 7.5 mg/kg intravenously on Day 1 of each 3-week treatment cycle. In addition, participants received capecitabine 1000 mg/m^2 orally twice daily on Days 1-14 of each 3-week treatment cycle.
  Interventions: Drug: Bevacizumab; Drug: Capecitabine
- Capecitabine (Active Comparator): Participants received capecitabine 1000 mg/m^2 orally twice daily on Days 1-14 of each 3-week treatment cycle.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Bevacizumab — Treatment continued until unacceptable toxicity, withdrawal of consent, disease progression, or a decision to terminate at the discretion of the Investigator if medically indicated. Bevacizumab was supplied in single-use vials.
  Other Names: Avastin
  Arms: Bevacizumab + capecitabine
Drug: Capecitabine — Treatment continued until unacceptable toxicity, withdrawal of consent, disease progression, or a decision to terminate at the discretion of the Investigator if medically indicated. Capecitabine was supplied as tablets.
  Other Names: Xeloda

SUMMARY:
This 2-arm study assessed the efficacy and safety of bevacizumab (Avastin) in combination with capecitabine (Xeloda), compared with capecitabine alone, in elderly patients with metastatic colorectal cancer. Patients were randomized to receive either bevacizumab (7.5 mg/kg intravenously on Day 1 of each 3-week cycle) in combination with capecitabine (1000 mg/m^2 orally twice a day on Days 1-14 of each 3-week cycle) or capecitabine (1000 mg/m^2 orally twice a day on Days 1-14 of each 3-week cycle) alone.

No notable trends or interactions in laboratory values, electrocardiogram, or vital signs suggesting an effect in either direction for capecitabine/bevacizumab combination therapy or capecitabine monotherapy were observed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥ 70 years of age.
* Cancer of the colon or rectum.
* Metastatic disease diagnosed ≤ 6 months before enrollment.
* ≥ 1 measurable metastatic lesion.

Exclusion Criteria:

* Adjuvant anti-vascular endothelial growth factor (VEGF) treatment.
* Prior chemotherapeutic treatment for metastatic colorectal cancer.
* Past or current history of other malignancies (with the exception of basal and squamous cell cancer of the skin, or in situ cancer of the cervix).
* Clinically significant cardiovascular disease.
* Current or recent daily use of aspirin (> 325 mg/day) or other non-steroidal anti-inflammatory drug (NSAID), or full dose anticoagulants.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 280 (Actual)
Dates: Start 2007-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (48):
- Austria (4):
  - Innsbruck
  - Linz
  - Salzburg
  - Vienna
- Canada (7):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Greece (2):
  - Larissa
  - Piraeus
- Hungary (3):
  - Budapest
  - Győr
  - Zalaegerszeg-Pozva
- Italy (4):
  - Lecce, Apulia
  - Reggio Emilia, Emilia-Romagna
  - Rome, Lazio
  - Florence, Tuscany
- Mexico (3):
  - León
  - Mexico City
  - Puebla City
- Netherlands (3):
  - Apeldoorn
  - Eindhoven
  - Utrecht
- Poland (2):
  - Krakow
  - Warsaw
- Ljubljana, Slovenia
- South Korea (3):
  - Gyeonggi-do
  - Incheon
  - Seoul
- Spain (7):
  - Barcelona, Barcelona
  - Jaén, Jaen
  - Las Palmas de Gran Canaria, Las Palmas
  - Leganés, Madrid
  - Madrid, Madrid
  - Murcia, Murcia
  - Zaragoza, Zaragoza
- United Kingdom (9):
  - Bristol
  - Colchester
  - Glasgow
  - Leicester
  - London
  - Manchester
  - Nottingham
  - Rhyl
  - Sutton

REFERENCES:
- [Derived] Cunningham D, Lang I, Marcuello E, Lorusso V, Ocvirk J, Shin DB, Jonker D, Osborne S, Andre N, Waterkamp D, Saunders MP; AVEX study investigators. Bevacizumab plus capecitabine versus capecitabine alone in elderly patients with previously untreated metastatic colorectal cancer (AVEX): an open-label, randomised phase 3 trial. Lancet Oncol. 2013 Oct;14(11):1077-1085. doi: 10.1016/S1470-2045(13)70154-2. Epub 2013 Sep 10. PMID 24028813

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab + Capecitabine | Capecitabine
Started | 140 | 140
Completed | 0 | 0
Not Completed | 140 | 140
Not completed — Death | 9 | 13
Not completed — Adverse Event | 22 | 12
Not completed — Patient Withdrew Consent | 19 | 10
Not completed — Protocol Violation | 3 | 3
Not completed — Lost to Follow-up | 0 | 3
Not completed — Discretion of Investigator or Sponsor | 7 | 3
Not completed — Disease progression | 67 | 88
Not completed — Screen Failure | 2 | 2
Not completed — Reason Not Specified | 11 | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All participants randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + Capecitabine | Capecitabine | Total
Number analyzed (Participants) | 140 | 140 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.1 (4.18) | 76.5 (3.91) | 76.3 (4.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 56 | 112
  Male | 84 | 84 | 168

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time in months from the date of randomization to the date of disease progression or death from any cause, whichever occurred first. All measurable lesions (maximum of 5 per organ and 10 in total, those with the longest diameter and suitability for accurate repeated measurements) were identified as target lesions (TL). A sum of the longest diameter for all TLs was calculated and reported as the baseline sum longest diameter (SLD). All other lesions were identified as non-TLs and recorded at baseline. PD was defined as ≥ 20% increase in the sum of the longest diameter of TLs, taking as reference the smallest SLD recorded since treatment started, the unequivocal progression of existing non-TLs, or the appearance of 1 or more new lesions.
Time Frame: Baseline to the end of the study (up to 5 years 8 months)
Population: Intent-to-treat population: All participants randomized into the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Capecitabine | Capecitabine
Number analyzed (Participants) | 140 | 140
Months | 9.1 [7.3 to 11.3] | 5.1 [4.3 to 6.3]
Statistical Analysis 1: Comparison: Bevacizumab + Capecitabine vs Capecitabine; Test type: Superiority or Other; p < 0.001, Log Rank

2. Secondary Outcome: Best Overall Response (BOR)
Description: BOR was defined as the best response (complete response [CR], partial response [PR], stable disease [SD], progressive disease [PD], not evaluable [NE], or not assessed [NA]) recorded from the start of study treatment until disease progression (PD) or death. CR was defined as the disappearance of all target (TL) and non-target lesions (non-TL). PR was defined as ≥ 30% decrease in the sum of the longest diameter (SLD) of TLs, taking as reference the baseline SLD, or the persistence of 1 or more non-TLs. For TLs, SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SLD since treatment started. For non-TLs, SD was defined as the persistence of 1 or more lesions. PD was defined as ≥ 20% increase in the sum of the longest diameter of TLs, taking as reference the smallest SLD recorded since treatment started, the unequivocal progression of existing non-TLs, or the appearance of 1 or more new lesions.
Time Frame: Baseline to the end of the study (up to 5 years 8 months)
Population: Intent-to-treat population: All participants randomized into the study. Only participants with a response were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bevacizumab + Capecitabine | Capecitabine
Number analyzed (Participants) | 140 | 140
Percentage of participants
  Complete Response | 2.9 [0.8 to 7.2] | 1.4 [0.2 to 5.1]
  Partial Response | 17.1 [11.3 to 24.4] | 8.6 [4.5 to 14.5]
  Stable Disease | 54.3 [45.7 to 62.7] | 48.6 [40.0 to 57.2]
  Progressive Disease | 10.0 [5.6 to 16.2] | 21.4 [14.9 to 29.2]
  Not assessed | 15.7 [10.1 to 22.8] | 20.0 [13.7 to 27.6]
Statistical Analysis 1: Comparison: Bevacizumab + Capecitabine vs Capecitabine; This statistical analysis compared the number of responders in the 2 treatment groups. A responder was defined as any participant with a best overall response of complete response or partial response. There were 28 responders in the bevacizumab + capecitabine group and 14 responders in the capecitabine group; Test type: Superiority or Other; p = 0.029, Fisher Exact

3. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time in months from the first confirmed complete response (CR) or partial response (PR) until disease progression or death from any cause, whichever occurred first. CR was defined as the disappearance of all target (TL) and non-target lesions (non-TL). PR was defined as ≥ 30% decrease in the sum of the longest diameter (SLD) of TLs, taking as reference the baseline SLD, or the persistence of 1 or more non-TLs.
Time Frame: Baseline to the end of the study (up to 5 years 8 months)
Population: Intent-to-treat population: All participants randomized into the study. Only participants with a complete response or partial response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Capecitabine | Capecitabine
Number analyzed (Participants) | 28 | 14
Months | 9.7 [8.3 to 10.9] | 9.4 [6.2 to 12.6]

4. Secondary Outcome: Time to Response
Description: Time to response was defined as the time in months from the date of first study treatment to the date of the first documentation of complete response (CR) or partial response (PR), whichever occurred first. CR was defined as the disappearance of all target (TL) and non-target lesions (non-TL). PR was defined as ≥ 30% decrease in the sum of the longest diameter (SLD) of TLs, taking as reference the baseline SLD, or the persistence of 1 or more non-TLs. Participants who did not have a confirmed response were censored at the date of the last evaluable tumor assessment, or if that was unavailable, at the date of the first dose of study medication.
Time Frame: Baseline to the end of the study (up to 5 years 8 months)
Population: Intent-to-treat population: All participants randomized into the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Capecitabine | Capecitabine
Number analyzed (Participants) | 140 | 140
Months | NA [NA to NA] — The median and the lower and upper limits of the 95% confidence interval could not be calculated due to insufficient data. | NA [30.4 to NA] — The median and the upper limit of the 95% confidence interval could not be calculated due to insufficient data.

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time in months from randomization to death from any cause.
Time Frame: Baseline to the end of the study (up to 5 years 8 months)
Population: Intent-to-treat population: All participants randomized into the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Capecitabine | Capecitabine
Number analyzed (Participants) | 140 | 140
Months | 20.7 [16.6 to 26.0] | 17.0 [12.9 to 22.0]
Statistical Analysis 1: Comparison: Bevacizumab + Capecitabine vs Capecitabine; Test type: Superiority or Other; p = 0.130, Log Rank

6. Secondary Outcome: Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: The ECOG performance status is a scale used to quantify cancer patients' general well-being and activities of daily life. The scale ranges from 0 to 5, with 0 denoting perfect health and 5 indicating death. The 6 categories are 0=Asymptomatic (Fully active, able to carry on all predisease activities without restriction), 1=Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature), 2=Symptomatic, < 50% in bed during the day (Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours), 3=Symptomatic, > 50% in bed, but not bedbound (Capable of only limited self-care, confined to bed or chair 50% or more of waking hours), 4=Bedbound (Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair), 5=Death. Reported is the percentage of participants in each of the 6 ECOG performance status categories.
Time Frame: Baseline to the Safety Follow-up which occurred 28 days after the last dose of treatment (up to 5 years 8 months).
Population: Intent-to-treat population: All participants randomized into the study.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab + Capecitabine | Capecitabine
Number analyzed (Participants) | 140 | 140
Percentage of participants
  Week 7 ECOG = 0 (n=117,110) | 50.4 | 34.5
  Week 7 ECOG = 1 | 47.0 | 58.2
  Week 7 ECOG = 2 | 1.7 | 5.5
  Week 7 ECOG = 3 | 0.9 | 1.8
  Week 7 ECOG = 4 | 0.0 | 0.0
  Week 7 ECOG = 5 | 0.0 | 0.0
  Week 16 ECOG = 0 (n=88,77) | 50.0 | 36.4
  Week 16 ECOG = 1 | 45.5 | 51.9
  Week 16 ECOG = 2 | 3.4 | 11.7
  Week 16 ECOG = 3 | 1.1 | 0.0
  Week 16 ECOG = 4 | 0.0 | 0.0
  Week 16 ECOG = 5 | 0.0 | 0.0
  Week 25 ECOG = 0 (n=66,42) | 43.9 | 45.2
  Week 25 ECOG = 1 | 48.5 | 45.2
  Week 25 ECOG = 2 | 6.1 | 9.5
  Week 25 ECOG = 3 | 1.5 | 0.0
  Week 25 ECOG = 4 | 0.0 | 0.0
  Week 25 ECOG = 5 | 0.0 | 0.0
  Week 34 ECOG = 0 (n=48,24) | 39.6 | 33.3
  Week 34 ECOG = 1 | 58.3 | 58.3
  Week 34 ECOG = 2 | 0.0 | 8.3
  Week 34 ECOG = 3 | 2.1 | 0.0
  Week 34 ECOG = 4 | 0.0 | 0.0
  Week 34 ECOG = 5 | 0.0 | 0.0
  Safety Follow-up ECOG = 0 (n=89,82) | 33.7 | 32.9
  Safety Follow-up ECOG = 1 | 47.2 | 45.1
  Safety Follow-up ECOG = 2 | 12.4 | 14.6
  Safety Follow-up ECOG = 3 | 6.7 | 4.9
  Safety Follow-up ECOG = 4 | 0.0 | 1.2
  Safety Follow-up ECOG = 5 | 0.0 | 1.2

7. Secondary Outcome: Percentage of Participants Requiring Additional Treatment for Malignancy
Description: Reported is the percentage of participants requiring additional treatment for malignancy in the survival follow-up period.
Time Frame: Baseline to the end of the study (up to 5 years 8 months)
Population: Intent-to-treat population: All participants randomized into the study.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab + Capecitabine | Capecitabine
Number analyzed (Participants) | 140 | 140
Percentage of participants | 50.7 | 49.3

8. Secondary Outcome: Duration of Follow-up
Description: Duration of follow-up is defined as the time in days from randomization until disease progression or death, or time to censoring for overall survival.
Time Frame: Baseline to the end of the study (up to 5 years 8 months)
Population: Intent-to-treat population: All participants randomized into the study.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Bevacizumab + Capecitabine | Capecitabine
Number analyzed (Participants) | 140 | 140
Days | 540.5 (423.52) | 479.2 (401.01)

9. Secondary Outcome: AEs, Laboratory Parameters, Vital Signs
Time Frame: Throughout study
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Safety population: All participants who had at least 1 dose of study medication.
Arm/Group | Bevacizumab + Capecitabine | Capecitabine
Serious Adverse Events (participants affected / at risk) | 40/134 | 42/136
Other Adverse Events (participants affected / at risk) | 129/134 | 130/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Capecitabine (N=134) | Capecitabine (N=136)
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Intestinal obstruction (Gastrointestinal disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 2 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Ascites (Gastrointestinal disorders) | 0 | 3
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 2
General physical health deterioration (General disorders) | 1 | 2
Pain (General disorders) | 1 | 1
Death (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Cellulitis gangrenous (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Amnesia (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1
Thrombosis (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 3
Circulatory collapse (Vascular disorders) | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Impacted fracture (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 2
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Bone operation (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Capecitabine (N=134) | Capecitabine (N=136)
Diarrhoea (Gastrointestinal disorders) | 54 | 48
Nausea (Gastrointestinal disorders) | 32 | 37
Abdominal pain (Gastrointestinal disorders) | 31 | 21
Vomiting (Gastrointestinal disorders) | 28 | 16
Constipation (Gastrointestinal disorders) | 25 | 19
Stomatitis (Gastrointestinal disorders) | 14 | 14
Abdominal pain upper (Gastrointestinal disorders) | 11 | 5
Dyspepsia (Gastrointestinal disorders) | 9 | 4
Fatigue (General disorders) | 32 | 37
Asthenia (General disorders) | 30 | 22
Pyrexia (General disorders) | 24 | 16
Mucosal inflammation (General disorders) | 20 | 11
Oedema peripheral (General disorders) | 11 | 17
Pain (General disorders) | 11 | 6
Palmar-Plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 66 | 54
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 11 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 4
Rash (Skin and subcutaneous tissue disorders) | 6 | 12
Lethargy (Nervous system disorders) | 12 | 15
Headache (Nervous system disorders) | 10 | 5
Dizziness (Nervous system disorders) | 9 | 17
Dysgeusia (Nervous system disorders) | 8 | 6
Paraesthesia (Nervous system disorders) | 8 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 23 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 13
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 38 | 31
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 4
Hypertension (Vascular disorders) | 22 | 6
Insomnia (Psychiatric disorders) | 7 | 7
Proteinuria (Renal and urinary disorders) | 10 | 1
Neutropenia (Blood and lymphatic system disorders) | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.